CLINICAL TRIAL: NCT04254796
Title: Neural Mechanisms of Meditation Training in Healthy and Depressed Adolescents: An MRI Connectome Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-29083; 5R25MH060482 (NIH); 1R61AT009864-01A1 (NIH)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TARA Training (Experimental): 12-week group TARA Training
  Interventions: Behavioral: Training for Awareness, Resilience, and Action (TARA)
- Control (No Intervention): Waitlist Control

INTERVENTIONS:
Behavioral: Training for Awareness, Resilience, and Action (TARA) — This will be a 12-week group meditation training - Training for Awareness, Resilience, and Action (TARA)
  Arms: TARA Training

SUMMARY:
The primary objective will be to study changes in putamen structural connectivity in healthy teens with meditation training. Hypothesis: Putamen structural node strength will increase in the training group compared to controls.

R61 Go/No-Go Criteria. Detect an effect size (a threshold of Cohen's d > 0.20) in changes of the primary mechanistic outcome (Putamen structural node strength) by the described meditation training in 100 healthy adolescents that are 14-18 years old and retain at least 80% of randomized participants for primary outcome measurement at the end of the study regardless of adherence to the intervention.

The secondary objective will be to study changes in emotional problems in healthy teens with meditation training. Hypothesis: There will be a significant decrease in emotional problems measured with the Strengths and Difficulties Questionnaire (SDQ) in the training group compared to controls.

Design and Outcomes: The current research study design will utilize an individually randomized group treatment, open-label, waitlist-controlled clinical trial to test the efficacy and safety of the investigator's innovative mindfulness meditation intervention (Training for Awareness Resilience and Action [TARA]) on the primary outcome (Putamen structural node strength) and secondary outcome (emotional problems measured with the Strengths and Difficulties Questionnaire [SDQ]) in healthy adolescents between the ages of 14 to 18 years old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male adolescents, 14-18 years old
* Fluency in English

Exclusion Criteria:

* Subjects younger or older than 14-18 years old.
* Subjects who are not healthy. Subjects who are taking any psychotropic medication.
* MRI contraindications (ferromagnetic objects on or inside the body, e.g., braces) and pregnancy.
* Not allowable: Current mindfulness training (e.g. MBSR, MBCT, DBT) and/or practice with a typically sitting meditation or yoga of 20 or more minutes two or more times per week within 60 days prior to study entry.
* Potential adolescent subjects with current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to the study requirements will be excluded and not allowed to enter the study.
* Potential subjects with an inability or unwillingness to give written informed assent or whose legal guardian/representative are unable or unwilling to give written informed consent will be excluded and not allowed to enter the study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Tymofiyeva, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tymofiyeva O, Sipes BS, Luks T, Hamlat EJ, Samson TE, Hoffmann TJ, Glidden DV, Jakary A, Li Y, Ngan T, Henje E, Yang TT. Interoceptive brain network mechanisms of mindfulness-based training in healthy adolescents. Front Psychol. 2024 Aug 13;15:1410319. doi: 10.3389/fpsyg.2024.1410319. eCollection 2024. PMID 39193038

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TARA Training | Control
Started | 50 | 50
Completed | 45 | 49
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TARA Training | Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.81 (1.37) | 16.04 (1.29) | 15.93 (1.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 22 | 21 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 5 | 16
  Not Hispanic or Latino | 38 | 44 | 82
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 3 | 4
  White | 25 | 28 | 53
  More than one race | 19 | 9 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in Putamen Node Strength
Description: Change in the Putamen node strength assessed using diffusion MRI.
  Node strengths are calculated as the sum of connection weights between the brain region of interest and all other nodes in the network.
  Higher values of node strength in general indicate stronger white matter connectivity between a specific brain region and the other regions, often caused by higher myelination. Higher values of change in node strength, similarly, indicate a higher level of structural network change occurred within the tissue.
Time Frame: Baseline/randomization and 12 weeks after baseline/randomization
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | TARA Training | Control
Number analyzed (Participants) | 45 | 49
unitless | 0.73 (4.07) | -0.42 (4.30)
Statistical Analysis 1: Comparison: TARA Training vs Control; The goal of the analysis was to measure the effect size of the change in the primary mechanistic outcome (Putamen structural node strength), with a Go/No-Go threshold of Cohen's d > 0.20; Test type: Other — Calculation of the effect size (Cohen's d); Cohen's d = 0.27, 95% CI 2-sided [-0.13 to 0.68]

2. Secondary Outcome: Change in Emotional Problems
Description: Change in the level of emotional problems measured with the Strengths and Difficulties Questionnaire (SDQ). The emotional problems scores have a possible range of 0 to 10. Higher scores represent higher levels of emotional problems.
Time Frame: Baseline/randomization and 12 weeks after baseline/randomization
Population: Note: 12 weeks after randomization, emotional problems measured with SDQ weren't acquired in one additional subject in the control group (resulting in 48 subjects with the secondary outcome measure in the control group). The study records contain Note to File, which states that the subject completed their second MRI, and the subject and their parent received an email containing a link to the study questionnaire but they never completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TARA Training | Control
Number analyzed (Participants) | 45 | 48
score on a scale | 2.12 (9.82) | 0.20 (7.15)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Solicited adverse events in TARA participants were captured as follows: (1) before each TARA session participants were asked through a questionnaire: "Has there been any significant unfavorable change in your mental or physical health since last class?"; (2) if the participant answered "yes" to this question, then a study staff member asked the participant for additional details regarding the participant's answer and this information was recorded in the Adverse Event form.
Arm/Group | TARA Training | Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TARA Training (N=50) | Control (N=50)
Suicidal ideation leading to hospitalization. (Psychiatric disorders) | 1 (1) | 0 (0) — Parent states that the cause was family-related problems and was in no way related to the TARA intervention (study records contain Note to File)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT04254796/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT04254796/ICF_001.pdf